CLINICAL TRIAL: NCT04234425
Title: A Trauma-Informed Approach for Positive Youth Development for Montana
Brief Title: A Trauma-Informed Approach for Positive Youth Development for Montana Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Lauren Davis, Assistant Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Davis01
Record Dates: First submitted 2020-01-14; First posted 2020-01-21 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Depression, Anxiety; Adolescent Behavior; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders; Adolescent Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): 18 high school students in a weight training class will be assigned to this experimental group and will receive the one-hour intervention twice weekly for 8 weeks.
  Interventions: Behavioral: Trauma-Informed Yoga

INTERVENTIONS:
Behavioral: Trauma-Informed Yoga — Trauma-Informed Yoga practice held within a high school weight training class

SUMMARY:
Given the prevalence of suicide and mental health issues in rural Montana, this project is intended to help mitigate stressors that may contribute to poor behavioral and mental health in high school-aged children. The immediate goal is to determine viability of a partnership with a rural southwestern Montana school and test the feasibility of a piloted implementation of a trauma-informed yoga intervention to address behavioral health outcomes and positive youth development.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in a specific weight training class at predetermined high school in rural Montana

Exclusion Criteria:

* Students not enrolled in a specific weight training class at predetermined high school in rural Montana

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Davis, Doctoral, Principal Investigator — Montana State University
Locations (1):
- Park High School, Livingston, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group
Started | 18
Midpoint-Week 4 | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: High school students in rural Montana
Arm/Group | Experimental Group
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (0.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Testing
Description: Students will provide a saliva sample in which cortisol levels will be analyzed through salivary assay kits (through Salimetrics.com). Samples will be collected on the first day of the intervention, halfway through the intervention, and on the last day of the intervention to determine if the intervention has improved stress levels (as indicated by a reduction in cortisol levels). A biostatistician will provide analysis and conclusion of these samples at the conclusion of the study.
Time Frame: Baseline and 4 weeks (Midpoint)
Population: 18 students in a weight training class in a rural Montana high school
Measure: Mean (Standard Deviation); unit: ug/dl
Groups:
- Experimental Group-Midpoint Data (4 Weeks): 18 high school students in a weight training class (one student less than baseline due to attrition)
- Experimental Group-Baseline Data: 18 high school students in a weight training class
Arm/Group | Experimental Group-Midpoint Data (4 Weeks) | Experimental Group-Baseline Data
Number analyzed (Participants) | 18 | 18
ug/dl | 0.245 (0.1356) | 0.3088 (0.1552)

2. Secondary Outcome: Generalized Anxiety Disorder-7 Anxiety Scale
Description: This 7 item questionnaire is based on a likert scale of 0 (not at all) to 3 (nearly every day) for items related to anxiety disorders. The lowest score is a zero and the maximum score is a 21. A reduction in score from pre- to post-assessment indicates an improvement in symptomology.
Time Frame: Baseline and 7 weeks after beginning of intervention
Population: High School Students in rural Montana
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group
Number analyzed (Participants) | 18
score on a scale
  Post Survey Results | 4.20 (5.36)
  Pre-Survey Results | 7.33 (5.44)
Statistical Analysis 1: Comparison: Experimental Group; Test type: Other — paired t test; p = .017, t-test, 2 sided; Mean Difference (Final Values) = 2.702, Standard Deviation 5.36

3. Secondary Outcome: Patient Health Questionnaire for Adolescents
Description: This 9 item questionnaire is designed to evaluate severity of depressive symptoms in adolescents. It is scored on a Likert scale from 0 (not at all) to 3 (nearly every day) on items linked to depression indicators. The minimum score is a 0 and the maximum score is a 27, and a reduction in score from pre- to post-assessment indicates an improvement in symptomology.
Time Frame: Baseline and 7 weeks after beginning of intervention
Population: high school students in rural Montana
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group
Number analyzed (Participants) | 18
score on a scale
  Post-Survey Results | 4.20 (7.06)
  Pre-Survey Results | 6.72 (4.42)
Statistical Analysis 1: Comparison: Experimental Group; Test type: Other — paired t test; p = .08, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.20, Standard Deviation 7.06

4. Secondary Outcome: Strengths and Difficulties Questionnaire for Ages 11-17 (Overall Score)
Description: This 25 item questionnaire is a brief emotional and behavioral scale for adolescents based on psychological attributes. Items are scored on a Likert scale from 0 (Not True) to 2 (Certainly True). The range in overall scores is 0-40. A reduction in score from pre- to post-assessment indicates an improvement in symptomology/outcomes.
Time Frame: Baseline and 7 weeks after beginning of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group
Number analyzed (Participants) | 18
score on a scale
  Post-Survey Overall Score | 20.47 (7.33)
  Pre-Survey Overall Score | 23.72 (7.48)
Statistical Analysis 1: Comparison: Experimental Group; Test type: Other — paired t test; p = .026, t-test, 2 sided; Mean Difference (Final Values) = 20.47, Standard Deviation 7.33

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: No adverse events occurred.
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04234425/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04234425/Prot_SAP_001.pdf